CLINICAL TRIAL: NCT06955936
Title: An Open Randomized Study on the Efficacy and Safety of Hemoadsorption With Efferon CT in Patients With Cardiogenic Shock Complicating Acute Myocardial Infarction
Brief Title: Efferon CT Hemoadsorption for Cardiogenic Shock in Acute Myocardial Infarction
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Efferon JSC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: efferon-ct-2025-01
Record Dates: First submitted 2025-04-25; First posted 2025-05-02 (Actual); Last update posted 2025-06-05 (Actual); Status verified 2025-04

CONDITIONS: Myocardial Infarction; Cardiogenic Shock
Keywords: Hemoadsorption; Extracorporeal therapy; Cytokine adsorption; Hemoperfusion
MeSH Terms: conditions — Myocardial Infarction; Shock, Cardiogenic

STUDY DESIGN:
Intervention Model Description: Allocation of patients into groups will be done by stratified 1:1 randomisation.
  Patients will be stratified into 2 groups based on the severity of cardiogenic shock according to the SCAI classification (stages B and C).
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Baseline therapy (No Intervention): Standard therapy (according to the clinical guidelines "Cardiogenic Shock (2025)" issued by the "Russian Federation of Anaesthesiologists and Reanimatologists").
- Basic therapy + Efferon CT (Experimental): Standard therapy supplemented with a single session of hemoadsorption using Efferon CT.
  Interventions: Device: Efferon CT

INTERVENTIONS:
Device: Efferon CT — Efferon CT (JSC Efferon, Moscow, RF) is a device for extracorporeal blood purification by direct hemoadsorption. Detoxification is carried out by sorption of cytokines and other products of endogenous intoxication with a molecular size of up to 55 kDa.
  The therapy will be performed once no later than 4 hours after the diagnosis of cardiogenic shock.
  The duration of hemoadsorption is from 4 to 12 hours. The rate of hemoadsorption is from 80 to 150 ml/min. Anticoagulation is systemic (heparin or sodium citrate).
  Arms: Basic therapy + Efferon CT

SUMMARY:
Cardiogenic shock is the most severe manifestation of acute heart failure and remains the leading cause of death in patients hospitalised with acute myocardial infarction.

Cardiogenic shock is a well-known and potent trigger of the immune response, ischemia/reperfusion organ damage, hemolysis and release of free hemoglobin. The activation of immune cells leads to the release of cytokines and inflammatory mediators such as IL-6, IL-8, activated complement and others. As a result of myocardial ischaemia and reperfusion injury, a multiorgan dysfunction syndrome may develop.

The Efferon CT hemoadsorption device effectively removes cytokines and other pro-inflammatory molecules (≤55 kDa). This study evaluates whether this blood-filtering therapy can prevent organ failure in acute myocardial infarction patients with cardiogenic shock by eliminating inflammation-inducing mediators.

DETAILED DESCRIPTION:
Cardiogenic shock (CS) is a state of acute critical tissue hypoperfusion caused by impaired myocardial contractility. It is one of the most serious complications of acute coronary syndrome (ACS), particularly acute myocardial infarction (AMI). Cardiogenic shock develops in approximately 30-40% of ACS patients, with a one-year mortality rate of 50-60%.

Despite advances in modern cardiology-including widespread use of timely revascularization, vasopressors, inotropic agents, and mechanical circulatory support-CS-related mortality remains unacceptably high. Efferent therapy, which modulates the homeostasis of biological fluids (e.g., blood) through physical and chemical methods (filtration, apheresis, sorption), represents a promising approach.

Recent studies on the hemoadsorbent CytoSorb in acute cardiac pathology demonstrated reductions in inflammatory markers (IL-6, lactate), improved hemodynamic stability, and lower 30-day ICU mortality (52% vs. 80% SOFA-predicted). These findings highlight the potential of cytokine adsorption to mitigate systemic inflammation in CS.

The Efferon CT hemoadsorption device, which effectively removes cytokines and other pro-inflammatory molecules (≤55 kDa), may improve outcomes by alleviating CS symptoms and preventing multiple organ dysfunction.

ELIGIBILITY:
Inclusion Criteria:

* Not more than 4 hours after diagnosis Cardiogenic shock complicating acute myocardial infarction
* Stages B - C of cardiogenic shock according to SCAI
* Patient condition allows treatment with Efferon® CT device for at least 4 hours
* SOFA score 12 or less

Exclusion Criteria:

* Broken-heart syndrome (takotsubo cardiomyopathy)
* Postcardiotomy cardiogenic shock
* Acute myocardial infarction within the last 4 weeks
* Myocarditis
* Cardiac trauma
* Charlson comorbidity index greater than 9 points
* Chronic kidney disease, stage 5 D (requiring continuous hemodialysis)
* Acute pulmonary embolism
* Acute cerebral circulatory collapse
* Transfusion reaction
* Patients on immunosuppressive therapy for cancer and autoimmune diseases
* Pregnancy
* Any other clinical condition of the patient that in the opinion of the investigator precludes inclusion in this study

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2025-04-29 (Actual); Primary Completion 2027-04-29 (Estimated); Study Completion 2027-07-31 (Estimated)

PRIMARY OUTCOMES:
Time to Resolution of Cardiogenic Shock (Days) | 1-7 days
  Time from randomization to sustained hemodynamic stabilization, defined as:
  Mean arterial pressure (MAP) ≥65 mmHg and Heart rate ≤110 bpm and Cessation of vasopressors/inotropes (e.g., norepinephrine, dopamine) and mechanical circulatory support (MCS). Persistence of all criteria for ≥4 consecutive hours

SECONDARY OUTCOMES:
Need for vasopressor support | 0-72 hours
  Need for vasopressors according to the VIS 2020 heart rate scale (Vasoactive inotropic score), measure every 12 hours. VIS is calculated as a weighted sum of all administered vasoactive inotropic agents.
Pulmonary oxygen metabolic function | 1-7 days
  Measuring PaO2 / FiO2 index every 24 hours
SOFA score | 1-7 days
  The SOFA (Sequential Organ Failure Assessment) index is equal to the sum of six indicators. The higher the score, the greater the insufficiency of the system being assessed. The higher the overall index, the greater the degree of multiorgan dysfunction. Violation of the function of each organ (system) is assessed separately in dynamics against the background of intensive therapy. With a score of no more than 12, multiple organ dysfunctions are assumed, 13-17 points indicate the transition of dysfunction to insufficiency, a score of about 24 indicates a high probability of death. The lower the SOFA index, the less pronounced organ failure and the better the patient's survival prognosis.
  Calculation every 24 hours.
Duration of ventilation | 1-7 days
  The time (hours) from the onset of hemoadsorption to the time of disconnection from the ventilator within 7 days or discharge from hospital or transfer from intensive care (if earlier than 7 days).
ICU length of stay | 1-7 days
  Time (days) from the start of hemoadsorption to transfer from the ICU within 7 days or hospital discharge (if earlier than day 7).
Hospital length of stay | 1-7 days
  Time (days) from the start of hemoadsorption to hospital discharge.
Incidence and severity of AKI | 1-7 days
  Frequency of AKI (AKI verified by KDIGO 2012 criteria) and duration (hours) of RRT in patients with AKI

CONTACTS AND LOCATIONS:
Overall Officials: Vyacheslav Ryabov, PhD, MD, Principal Investigator — Tomsk NRMC Cardiology Research Institute
Locations (1):
- Tomsk NRMC Cardiology Research Institute, Tomsk, Russia